CLINICAL TRIAL: NCT00243386
Title: Advate Antihemophilic Factor (Recombinant), Plasma/Albumin Free Method (ADVATE rAHF-PFM): A Phase 4 Study Comparing Two Prophylactic Regimens in Subjects With Severe or Moderately Severe Hemophilia A
Brief Title: Prophylaxis Study of Recombinant Factor VIII Manufactured Protein-Free (rAHF-PFM) in Patients With Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060201
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard prophylaxis
  Interventions: Drug: Antihemophilic factor, recombinant, manufactured protein-free
- 2 (Experimental): PK-driven prophylaxis
  Interventions: Drug: Antihemophilic factor, recombinant, manufactured protein-free

INTERVENTIONS:
Drug: Antihemophilic factor, recombinant, manufactured protein-free — Standard prophylaxis: 20-40 IU/kg every 48+/-6 hours, actual dose determined by investigator
  Arms: 1
Drug: Antihemophilic factor, recombinant, manufactured protein-free — PK-driven prophylaxis: 20-80 IU/kg every 72+/-6 hours, actual dose determined by Baxter using an algorithm and the patient´s pharmacokinetic data
  Arms: 2

SUMMARY:
The primary purpose of this randomized, two-arm parallel clinical study in 66 previously treated patients with severe or moderately severe hemophilia A is to compare the rate of bleeding episodes for standard prophylaxis (20-40 IU/kg every 48 ± 6 hours; actual dose determined by the investigator) with that of alternate prophylaxis (20-80 IU/kg every 72 + 6 hours; actual dose determined by Baxter utilizing an algorithm and the patient's pharmacokinetic data). The rates of bleeding episodes for the on-demand regimen and the prophylaxis regimens will also be compared for the cross-over portion of the study. Enrolled patients will be treated originally on demand for a period of 6 months and then they will be randomized into one of the prophylaxis arms. Prophylactic treatment will last for a period of 12 months +/- 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The subject has severe or moderately severe hemophilia A as defined by a baseline factor VIII level <= 2% of normal, as tested at screening
* The subject has a documented history of at least 150 exposure days to factor VIII concentrates (either plasma-derived or recombinant)
* The subject is within 7 to 65 years of age
* The subject has a Karnofsky performance score > (greater than) 60
* The subject is human immunodeficiency virus negative (HIV-) or is HIV+ with a CD4 count >= 400 cells/mm³ (CD4 count determined at screening, if necessary)
* The subject has been on a documented on-demand treatment regimen for at least 12 months immediately prior to enrollment
* The subject has a documented history (e.g. in medical charts or dispensing information, or signed investigator statement) of at least 8 joint hemorrhages in the 12 months immediately prior to enrollment
* The subject resides within the coverage area of the mobile compliance device; coverage area will be determined at screening
* The subject or the subject's legally authorized representative has provided written informed consent

Exclusion Criteria:

* The subject has a known hypersensitivity to factor VIII concentrates or mouse or hamster proteins
* The subject has a history of factor VIII inhibitors with a titer >= 0.6 BU (by Bethesda or Nijmegen assay) at any time prior to screening
* The subject has a detectable factor VIII inhibitor at screening, with a titer >= 0.4 BU (by Nijmegen Assay) in the central laboratory
* The subject has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) > 1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.
* The subject has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (e.g., qualitative platelet defect or von Willebrand's Disease)
* The subject has been treated during the last sixty (60) days prior to or is being treated at screening/enrollment with an immunomodulating drug.
* The subject has participated in another investigational study within thirty (30) days of enrollment
* The subject has previously participated in a clinical study with rAHF-PFM
* The subject's clinical condition may require a major surgery (defined as moderate to critical risk and perioperative blood loss ≥ 500 mL) during the period of the subject's participation in the study
* The subject is female of childbearing potential with a positive pregnancy test

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-01-04 (Actual); Primary Completion 2010-06-16 (Actual); Study Completion 2010-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (29):
- United States (9):
  - Los Angeles, California
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Minneapolis, Minnesota
  - New York, New York
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Seattle, Washington
- Vienna, Austria
- Czechia (2):
  - Brno
  - Prague
- Athens, Greece
- Hungary (5):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
  - Szombathely
- Italy (2):
  - Florence
  - Milan
- Poland (5):
  - Gdansk
  - Krakow
  - Lublin
  - Warsaw
  - Wroclaw
- Moscow, Russia
- Ljubljana, Slovenia
- United Kingdom (2):
  - Cardiff
  - Nottingham

REFERENCES:
- [Derived] Valentino LA, Mamonov V, Hellmann A, Quon DV, Chybicka A, Schroth P, Patrone L, Wong WY; Prophylaxis Study Group. A randomized comparison of two prophylaxis regimens and a paired comparison of on-demand and prophylaxis treatments in hemophilia A management. J Thromb Haemost. 2012 Mar;10(3):359-67. doi: 10.1111/j.1538-7836.2011.04611.x. PMID 22212248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 21 European and 9 United States clinical sites beginning January 2006 and completing in June 2010
Pre-assignment Details: 82 participants were enrolled and screened. 7 were screen failures, 1 was withdrawn for non-compliance, and 1 requested withdrawal. Therefore, 73 of the 82 enrolled were exposed to investigational product in the first part of the study (on-demand treatment).
Groups:
- All Study Participants: Participants first underwent an open-label pharmacokinetic (PK) evaluation of rAHF-PFM. 48 hours after the initial PK study, a 6 month period of on-demand treatment was conducted (Part 1). After completing the on-demand treatment, participants were randomized to 1 of 2 prophylactic regimens for 12 months ±2 weeks (Part 2). The standard prophylactic regimen was dosed at 20 to 40 IU/kg every 48 ±6 hours, and the PK-driven prophylaxis regimen was dosed at 20 to 80 IU/kg every 72 ±6 hours.
- PK-Driven Prophylaxis: The PK-driven prophylaxis regimen was dosed at 20 to 80 IU/kg of rAHF-PFM every 72 ±6 hours
- Standard Prophylaxis: The standard prophylactic regimen was dosed at 20 to 40 IU/kg of rAHF-PFM every 48 ±6 hours
Period: On-Demand Regimen (Study Part 1)
Arm/Group | All Study Participants | PK-Driven Prophylaxis | Standard Prophylaxis
Started | 73 | 0 (Participants were randomized to PK-Driven or Standard Prophylaxis after Part 1 (On-Demand Regimen)) | 0 (Participants were randomized to PK-Driven or Standard Prophylaxis after Part 1 (On-Demand Regimen))
Completed | 69 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Screen Failures | 2 | 0 | 0
Period: End of Part 1, But Prior to Prophylaxis
Arm/Group | All Study Participants | PK-Driven Prophylaxis | Standard Prophylaxis
Started | 69 | 0 (Participants were randomized to PK-Driven or Standard Prophylaxis after Part 1 (On-Demand Regimen)) | 0 (Participants were randomized to PK-Driven or Standard Prophylaxis after Part 1 (On-Demand Regimen))
Completed | 66 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawn for Non-Compliance | 1 | 0 | 0
Period: PK-Driven or Standard Prophylaxis
Arm/Group | All Study Participants | PK-Driven Prophylaxis | Standard Prophylaxis
Started | 0 (Participants were randomized to PK-Driven or Standard Prophylaxis after Part 1 (On-Demand Regimen)) | 34 | 32
Completed | 0 | 31 | 32
Not Completed | 0 | 3 | 0
Not completed — Withdrawn for Non-Compliance | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants first underwent an open-label evaluation of rAHF-PFM PK. 48 hours after the initial PK study, a 6 month period of on-demand treatment was conducted (Part 1). After completing the on-demand treatment, participants were randomized to 1 of 2 prophylactic regimens for 12 months ±2 weeks (Part 2). The standard prophylactic regimen was dosed at 20 to 40 IU/kg every 48 ±6 hours, and the PK-driven prophylaxis regimen was dosed at 20 to 80 IU/kg every 72 ±6 hours.
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
Age, Continuous [Median (Full Range); unit: years] | 26 [7 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Mean Transformed Annualized Bleed Rate Estimates From Each of the 1-year Prophylaxis Regimens
Description: Participants were Randomized to Receive 1 of the 2 Following Prophylaxis Regimens (Study Part 2): 1. Standard prophylaxis (20-40 IU/kg (every 48 ±6 hour), exact regimen determined by investigator) 2. PK-driven prophylaxis (20-80 IU/kg (every 72 ±6 hour), exact regimen determined by sponsor) Annualized bleed rates were transformed using the square root of the number of bleeding episodes observed (X = bleeds/year), X' = √(X + 0.5). This transformation was performed to stabilize the variance and align the sample distribution with the assumption of normality inherent in using the t-test.
Time Frame: 12 months ±2 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: (bleeds/year)^(1/2)
Groups:
- PK-Driven Prophylaxis: PK-driven prophylaxis regimen dosed at 20 to 80 IU/kg every 72 ±6 hours
- Standard Prophylaxis: Standard prophylaxis regimen dosed at 20 to 40 IU/kg every 48 ±6 hours
Arm/Group | PK-Driven Prophylaxis | Standard Prophylaxis
Number analyzed (Participants) | 23 | 30
(bleeds/year)^(1/2) | 1.61 (1.10) | 1.46 (0.98)
Statistical Analysis 1: Comparison: PK-Driven Prophylaxis vs Standard Prophylaxis; A t-test was used to compare the means of the transformed data. The null-hypothesis tested was H0: X'A(PK-driven prophylaxis) - X'B (standard prophylaxis) = 0 (i.e., no difference for treatment under the 2 prophylactic regimens. X' = (ABR+0.5)^(1/2); Test type: Superiority or Other; p = 0.6016, t-test, 2 sided

2. Secondary Outcome: Mean Difference of Transformed Annualized Bleeding Rate Between On-Demand and Standard Prophylaxis Treatment Regimens
Description: Annualized bleed rates were transformed using the square root of the number of bleeding episodes observed (X bleeds/year), X' = √(X + 0.5). This transformation was performed to stabilize the variance and align the sample distribution with the assumption of normality inherent in using the paired t-test. Mean Difference of Transformed Annualized Bleeding Rate (TABR) = (On-Demand Treatment TABR) - (Standard Prophylaxis Treatment TABR). Participants from the On-Demand portion of the study were subsequently randomized to either Standard Prophylaxis or PK-Driven Prophylaxis, (i.e the same participants were analyzed across the two measurement time periods).
Time Frame: On-demand 6 months (± 2 weeks); followed by Prophylaxis 12 months (± 2 weeks)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: (bleeds/year)^(1/2)
Groups:
- On-Demand Versus Standard Prophylaxis: On-demand: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, Gastrointestinal (GI), and intracranial (60-100 IU/kg every 8-12 hours) Standard Prophylaxis: 20-40 IU/kg (every 48 ± 6 hours), exact regimen to be determined by the investigator
Arm/Group | On-Demand Versus Standard Prophylaxis
Number analyzed (Participants) | 32
(bleeds/year)^(1/2) | 5.29 (1.46)
Statistical Analysis 1: Comparison: On-Demand Versus Standard Prophylaxis; Test type: Superiority or Other; p < 0.0001, Paired t-Test — 2-sided paired T-tests were done comparing transformed annualized bleeding rates between On-Demand and Prophylaxis regimens

3. Secondary Outcome: Mean Difference of Transformed Annualized Bleeding Rate Between On-Demand and PK-Driven Prophylaxis Treatment Regimens
Description: Annualized bleed rates were transformed using the square root of the number of bleeding episodes observed (X bleeds/year), X' = √(X + 0.5). This transformation was performed to stabilize the variance and align the sample distribution with the assumption of normality inherent in using the paired t-test. Mean Difference of Transformed Annualized Bleeding Rate (TABR) = (On-Demand Treatment TABR) - (PK-Driven Prophylaxis Treatment TABR) Participants from the On-Demand portion of the study were subsequently randomized to either Standard Prophylaxis or PK-Driven Prophylaxis, (i.e the same participants were analyzed across the two measurement time periods).
Time Frame: On-demand 6 months (± 2 weeks); followed by Prophylaxis 12 months (± 2 weeks)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: (bleeds/year)^(1/2)
Groups:
- On-Demand Versus PK-Driven Prophylaxis: On-demand: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours) PK-driven prophylaxis: 20-80 IU/kg (every 72 ± 6 hours), exact regimen to be determined by the sponsor
Arm/Group | On-Demand Versus PK-Driven Prophylaxis
Number analyzed (Participants) | 34
(bleeds/year)^(1/2) | 5.00 (1.85)
Statistical Analysis 1: Comparison: On-Demand Versus PK-Driven Prophylaxis; Test type: Superiority or Other; p < 0.0001, Paired t-test — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Mean Difference of Transformed Annualized Bleeding Rate Between On-Demand and Any Prophylaxis Treatment Regimens
Description: Annualized bleed rates were transformed using the square root of the number of bleeding episodes observed (X bleeds/year), X' = √(X + 0.5). This transformation was performed to stabilize the variance and align the sample distribution with the assumption of normality inherent in using the paired t-test. Mean Difference of Transformed Annualized Bleeding Rate (TABR) = (On-Demand Treatment TABR) - (Any Prophylaxis Treatment TABR). Any Prophylaxis = Standard or PK-Driven Prophylaxis Participants from the On-Demand portion of the study were subsequently randomized to either Standard Prophylaxis or PK-Driven Prophylaxis, (i.e the same participants were analyzed across the two measurement time periods).
Time Frame: On-demand 6 months (± 2 weeks); Prophylaxis 12 months (± 2 weeks)
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: (bleeds/year)^(1/2)
Groups:
- On-Demand Versus Any Prophylaxis: On-demand: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours) Prophylaxis: •Standard prophylaxis: 20-40 IU/kg (every 48 ± 6 hours), exact regimen to be determined by the investigator •PK-driven prophylaxis: 20-80 IU/kg (every 72 ± 6 hours), exact regimen to be determined by the sponsor
Arm/Group | On-Demand Versus Any Prophylaxis
Number analyzed (Participants) | 66
(bleeds/year)^(1/2) | 5.14 (1.66)
Statistical Analysis 1: Comparison: On-Demand Versus Any Prophylaxis; Test type: Superiority or Other; p < 0.0001, Paired t-test — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Total Weight-Adjusted Dose of rAHF-PFM Used Per Year for Each Prophylaxis Arm
Description: Participants were Randomized to Receive 1 of the 2 Following Prophylaxis Regimens (Part 2 of the study): 1. Standard prophylaxis- infusions every 48 ±6 hours, dosed at 20 to 40 IU/kg. 2. PK-driven prophylaxis- infusions every 72 ±6 hours dosed at 20 to 80 IU/kg.
Time Frame: 12 months ±2 weeks
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: IU/kg
Arm/Group | PK-Driven Prophylaxis | Standard Prophylaxis
Number analyzed (Participants) | 34 | 32
IU/kg | 5197.8 [3268.4 to 8273.5] | 5768.2 [4728.0 to 6425.4]
Statistical Analysis 1: Comparison: PK-Driven Prophylaxis vs Standard Prophylaxis; Test type: Superiority or Other; p = 0.4924, Wilcoxon-Rank Sum (Mann-Whitney)

6. Secondary Outcome: Bleeding Episodes Treated With 1 to ≥4 Infusions
Description: The number of bleeding episodes treated with 1, 2, 3, or ≥4 infusions of rAHF-PFM to achieve adequate hemostasis
Time Frame: Throughout the study period (4 years and 5 months)
Population: Intent to Treat Efficacy Set
Measure: Number; unit: Bleeding episodes
Groups:
- On-Demand Treatment: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours)
- Standard Prophylaxis Treatment: 20-40 IU/kg (every 48 ± 6 hours), exact regimen to be determined by the investigator
- PK-Driven Prophylaxis: 20-80 IU/kg (every 72 ± 6 hours), exact regimen to be determined by the sponsor
Arm/Group | On-Demand Treatment | Standard Prophylaxis Treatment | PK-Driven Prophylaxis
Number analyzed (Participants) | 62 | 13 | 22
Bleeding episodes
  1 infusion (n = 62, 13, 22) | 1168 | 68 | 90
  2 infusions (n = 51, 6, 9) | 277 | 12 | 37
  3 infusions (n = 27, 2, 4) | 128 | 4 | 5
  4 or more infusions (n = 21, 5, 5) | 50 | 9 | 7

7. Secondary Outcome: Assessment of Hemostasis for Treatment of Bleeding Episodes
Description: Number of rAHF-PFM-treated bleeding episodes with an assessment of hemostasis (4-point ordinal scale): Excellent: Full pain relief & bleeding cessation within ~8 hrs of 1 infusion. Additional infusions may have been given to maintain hemostasis; Good: Definite pain relief and/or improvement in bleeding within ~8 hrs after infusion. Possibly requires >1 infusion for complete resolution; Fair: Probable or slight relief of pain & slight improvement in bleeding within ~8 hrs after infusion. Requires >1 infusion for complete resolution; None: No improvement or condition worsens
Time Frame: On-demand 6 months (± 2 weeks); Prophylaxis 12 months (± 2 weeks)
Population: Hemostatic Efficacy Rating Analysis Set (Participants with bleeding episodes that were rated)
Measure: Number; unit: bleeding episodes
Groups:
- On-Demand Regimen: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours)
- Standard Prophylaxis: 20-40 IU/kg (every 48 ± 6 hours), exact regimen to be determined by the investigator
Arm/Group | On-Demand Regimen | Standard Prophylaxis | PK-Driven Prophylaxis
Number analyzed (Participants) | 70 | 18 | 25
bleeding episodes
  Excellent | 547 | 39 | 33
  Good | 943 | 38 | 75
  Fair | 167 | 16 | 11
  None | 3 | 0 | 20
  Unknown | 13 | 0 | 0

8. Secondary Outcome: Total Area Under the Curve (AUC)
Description: Total AUC estimated by AUC 0-48h plus an area extrapolated from the log-linear regression model
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
IU*h/dL | 1334.45 (454.33) | 1061.26 (452.87)

9. Secondary Outcome: Area Under the Curve
Description: Area under the factor VIII (FVIII) plasma concentration versus time curve (AUC) from 0 to 48 hours estimated using the linear trapezoidal method
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
IU*h/dL | 1213.98 (323.96) | 966.68 (330.83)

10. Secondary Outcome: Maximum Plasma Concentration (C-max)
Description: Maximal Factor VIII Concentration After Infusion
Time Frame: Within 1 hour post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: IU/dL
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
IU/dL | 91.12 (20.15) | 74.47 (11.30)

11. Secondary Outcome: Adjusted Incremental Recovery (IR)
Description: Change in factor VIII concentration from pre- to post-infusion at initial and termination study visits. Adjusted IR defined as: [Cmax (IU/dL) - pre-infusion FVIII (IU/dL)]/dose (IU/kg)
Time Frame: 30 minutes pre-infusion to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Geometric Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
IU/dL per IU/kg | 1.81 (0.41) | 1.47 (0.27)

12. Secondary Outcome: Terminal Half-life
Description: Computed from the regression slope in the terminal phase of the model. Terminal half life is the time it takes for the plasma concentration or the amount of drug in the body to be reduced by 50%.
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
hours | 13.91 (5.07) | 14.66 (5.21)

13. Secondary Outcome: Weight-Adjusted Clearance
Description: Computed as the weight-adjusted dose divided by total AUC
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: mL/(kg*h)
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
mL/(kg*h) | 3.89 (1.21) | 5.17 (1.94)

14. Secondary Outcome: Mean Residence Time
Description: Computed as total Area Under the Moment Curve (AUMC) divided by the total AUC
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
hours | 17.71 (7.16) | 17.88 (5.67)

15. Secondary Outcome: Volume of Distribution at Steady State
Description: Computed as weight-adjusted clearance * mean residence time
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Intent to Treat Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | ≥14 Years of Age | <14 Years of Age
Number analyzed (Participants) | 65 | 6
dL/kg | 0.65 (0.19) | 0.84 (0.19)

16. Secondary Outcome: Factor VIII Inhibitor Development
Description: Number of treated participants who developed factor VIII inhibitors
Time Frame: Throughout study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: Participants
Groups:
- All Study Participants: All participants who were exposed to Investigational Product (IP)
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
Participants | 0

17. Secondary Outcome: Number of Participants With AEs Related to Investigational Product (IP)
Description: Number of treated participants with AEs judged to be possibly or probably related to treatment with IP
Time Frame: Throughout study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: Participants
Groups:
- All Study Participants: All participants who were exposed to IP
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
Participants | 4

18. Secondary Outcome: Number of Participants Who Reported ≥1 AE Regardless of Relatedness to Investigational Product (IP)
Description: Number of treated participants with 1 or more AE regardless of relatedness to IP
Time Frame: Throughout study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
Participants | 44

19. Secondary Outcome: Number of Participants Who Reported ≥1 AE Regardless of Relatedness to IP by Treatment Regimen
Time Frame: Throughout the study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- On-Demand: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours)
Arm/Group | On-Demand | Standard Prophylaxis | PK-Driven Prophylaxis
Number analyzed (Participants) | 72 | 32 | 34
participants | 33 | 15 | 19

20. Secondary Outcome: Number of Participants With SAEs by Preferred MedDRA Term and Treatment Regimen
Time Frame: Throughout the study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- SAEs Outside of the 3 Treatment Arms: Participants with SAEs that occurred after exposure to investigational product, but outside of the three treatment arms
Arm/Group | On-Demand | Standard Prophylaxis | PK-Driven Prophylaxis | SAEs Outside of the 3 Treatment Arms
Number analyzed (Participants) | 72 | 32 | 34 | 1
participants
  ABDOMINAL PAIN | 1 | 0 | 0 | 0
  NAUSEA | 1 | 0 | 0 | 0
  TOOTH ABSCESS | 1 | 0 | 0 | 0
  JOINT DISLOCATION | 1 | 0 | 0 | 0
  HAEMOPHILIC ARTHROPATHY | 1 | 0 | 1 | 0
  SYNOVITIS | 1 | 0 | 0 | 0
  CALCULUS URINARY | 1 | 0 | 0 | 0
  HOSPITALIZATION | 1 | 0 | 0 | 0
  PULPITIS DENTAL | 0 | 1 | 0 | 0
  SOMNAMBULISM | 0 | 1 | 0 | 0
  FACTOR VIII INHIBITION (UNCONFIRMED) | 0 | 0 | 1 | 0
  APPENDICITIS | 0 | 0 | 1 | 0
  PAIN IN EXTREMITY | 0 | 0 | 0 | 1

21. Secondary Outcome: AEs With Onset ≤1 Hour Following the End of an Infusion, Regardless of Relatedness
Time Frame: Throughout study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: Events
Arm/Group | All Study Participants
Number analyzed (Participants) | 73
Events | 39

22. Secondary Outcome: Number of Participants With Severe SAEs and Severe Non-SAEs by Preferred MedDRA Term and Treatment Regimen
Description: This outcome is focused only on SEVERE SAEs and SEVERE non-SAEs
Time Frame: Throughout the study period (4 years and 5 months)
Population: Safety Analysis Set
Measure: Number; unit: participants
Groups:
- On-Demand: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours
Arm/Group | On-Demand | Standard Prophylaxis | PK-Driven Prophylaxis
Number analyzed (Participants) | 72 | 32 | 34
participants
  TOOTH ABSCESS (SAE) | 1 | 0 | 0
  HAEMOPHILIC ARTHROPATHY (SAE) | 0 | 0 | 1
  HAEMOPHILIC ARTHROPATHY (non-SAE) | 1 | 0 | 1
  ABDOMINAL PAIN (non-SAE) | 1 | 0 | 0
  ARTHRALGIA (non-SAE) | 1 | 0 | 0

23. Secondary Outcome: Baseline Health-related Quality of Life (HRQoL) Scores: PF, RP, BP, GH, VT, SF, RE, MH, PCS, and MCS
Description: Physical Functioning (PF); Role Limitation Due to Physical Health (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role Limitation Due to Emotional Problems (RE); Mental Health (MH), Physical Component Score (PCS); Mental Component Score (MCS). Baseline SF-36v1 Scores, where data available. Scores range 0-100, higher scores represent better health. There is no total overall score; scoring is done for subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores.
Time Frame: Baseline
Population: Safety Analysis Set
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Assessed Before Treatment
Number analyzed (Participants) | 71
Scores on a scale
  Physical Functioning (PF) | 44.56 [17.29 to 57.14]
  Role-Physical (RP) | 42.10 [27.95 to 56.24]
  Bodily Pain (BP) | 46.48 [25.07 to 62.75]
  General Health (GH) | 43.87 [19.52 to 64.00]
  Vitality (VT) | 51.42 [25.39 to 67.20]
  Social Functioning (SF) | 46.28 [19.14 to 57.14]
  Role-Emotional (RE) | 55.34 [23.74 to 55.34]
  Mental Health (MH) | 50.44 [20.91 to 64.07]
  Physical Component Score (PCS) | 42.32 [20.10 to 67.67]
  Mental Component Score (MCS) | 52.65 [22.56 to 68.10]

24. Secondary Outcome: Health-related Quality of Life (HRQoL) Scores: PF, RP, BP, GH, VT, SF, RE, MH, PCS, and MCS at the End of Treatment Regimens
Description: as for outcome 23
Time Frame: End of on-demand treatment period (6 months) and at study termination (approximately 18 months)
Population: Pharmacoeconomic Analysis Set
Measure: Median (Full Range); unit: Scores on a scale
Groups:
- On-Demand Treatment: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours
- Any Prophylaxis Treatment: Any Prophylaxis Treatment (either Standard Prophylaxis or PK-Driven Prophylaxis) Standard Prophylaxis: 20-40 IU/kg (every 48 ± 6 hours), exact regimen to be determined by the investigator PK-Driven Prophylaxis: 20-80 IU/kg (every 72 ± 6 hours), exact regimen to be determined by the sponsor
Arm/Group | On-Demand Treatment | Standard Prophylaxis | PK-Driven Prophylaxis | Any Prophylaxis Treatment
Number analyzed (Participants) | 63 | 31 | 34 | 65
Scores on a scale
  Bodily Pain (BP) | 46.5 [29.4 to 62.8] | 51.6 [19.9 to 62.8] | 51.6 [29.4 to 62.8] | 51.6 [19.9 to 62.8]
  General Health (GH) | 43.9 [19.5 to 64.0] | 48.6 [19.5 to 64.0] | 46.2 [29.8 to 60.3] | 48.6 [19.5 to 64.0]
  Mental Component Score (MCS), On-Demand n=62 | 54.9 [22.8 to 69.9] | 56.1 [13.3 to 69.6] | 54.5 [11.4 to 62.5] | 55.0 [11.4 to 69.6]
  Mental Health (MH), On-Demand n=62 | 51.6 [14.1 to 64.1] | 50.4 [20.9 to 64.1] | 52.7 [7.3 to 64.1] | 50.4 [7.3 to 64.1]
  Physical Component Score (PCS), On-Demand n=62 | 44.0 [16.1 to 61.2] | 50.2 [17.6 to 68.8] | 47.3 [25.3 to 62.3] | 47.8 [17.6 to 68.8]
  Physical Functioning (PF), On-Demand n=62 | 48.8 [17.3 to 57.1] | 46.7 [21.5 to 57.1] | 46.7 [17.3 to 57.1] | 46.7 [17.3 to 57.1]
  Role Emotional (RE) | 55.3 [23.7 to 55.3] | 55.3 [23.7 to 55.3] | 55.3 [23.7 to 55.3] | 55.3 [23.7 to 55.3]
  Role Physical (RP) | 49.2 [28.0 to 56.2] | 56.2 [28.0 to 56.2] | 56.2 [28.0 to 56.2] | 56.2 [28.0 to 56.2]
  Social Functioning (SF) | 46.3 [30.0 to 57.1] | 51.7 [24.6 to 57.1] | 51.7 [13.7 to 57.1] | 51.7 [13.7 to 57.1]
  Vitality (VT) | 53.8 [32.5 to 70.4] | 56.2 [27.8 to 70.4] | 56.2 [23.0 to 68.0] | 56.2 [23.0 to 70.4]

25. Secondary Outcome: HRQoL Scores Change From On-Demand Treatment Regimen Period Through Prophylaxis Period
Description: Differences in health domain scores = (End of on-demand treatment) - (End of prophylaxis regimen). A negative value for the median difference equates to a larger domain score for the prophylaxis regimen Physical Functioning (PF); Role Limitation Due to Physical Health (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role Limitation Due to Emotional Problems (RE); Mental Health (MH), Physical Component Score (PCS); Mental Component Score (MCS). Scores range 0-100, higher scores represent better health. There is no total overall score; scoring is done for subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores for each of the 8 HRQoL/SF-36 health domain scores.
Time Frame: End of on-demand treatment period (6 months) and at study termination (approximately 18 months)
Population: Pharmacoeconomic Analysis Set ≥14 Years and Older
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | On-Demand to Standard Prophylaxis | On-Demand to PK-Driven Prophylaxis | On-Demand to Any Prophylaxis Treatment
Number analyzed (Participants) | 27 | 30 | 57
Scores on a scale
  Physical Functioning (PF) | 0.00 [-10.48 to 14.68] | -2.10 [-18.88 to 20.97] | -2.10 [-18.88 to 20.97]
  Role Physical (RP) | 0.00 [-28.29 to 21.21] | 0.00 [-28.29 to 28.29] | 0.00 [-28.29 to 28.29]
  Bodily Pain (BP) | 0.00 [-29.55 to 17.55] | -4.29 [-25.27 to 13.28] | 0.00 [-29.55 to 17.55]
  General Health (GH) | -3.74 [-29.55 to 17.55] | -2.34 [-21.07 to 18.73] | -2.34 [-20.13 to 17.79]
  Vitality (VT) | 0.00 [-9.47 to 23.67] | 0.00 [-16.57 to 30.77] | 0.00 [-16.57 to 30.77]
  Social Functioning (SF) | 0.00 [-21.72 to 16.29] | 0.00 [-16.29 to 16.29] | 0.00 [-21.72 to 16.29]
  Role Emotional (RE) | 0.00 [-10.53 to 31.60] | 0.00 [-31.60 to 21.07] | 0.00 [-31.60 to 31.60]
  Mental Health (MH) | 0.00 [-13.63 to 15.90] | -1.13 [-40.90 to 34.08] | 0.00 [-40.90 to 34.08]
  Physical Component Score (PCS) | -2.55 [-20.22 to 8.69] | -3.14 [-16.78 to 19.70] | -2.76 [-20.22 to 19.70]
  Mental Component Score (MCS) | 1.52 [-8.31 to 21.64] | 0.79 [-35.25 to 24.56] | 1.30 [-35.25 to 24.56]

26. Primary Outcome: Median Annualized Bleed Rate Estimates From Each of the 1 Year Prophylaxis Regimens
Description: as for outcome 5
Time Frame: 12 months ±2 weeks
Population: Intent to treat
Measure: Median (Full Range); unit: Bleeds per year
Arm/Group | PK-Driven Prophylaxis | Standard Prophylaxis
Number analyzed (Participants) | 34 | 32
Bleeds per year | 2.01 [0.00 to 17.06] | 1.00 [0.00 to 25.87]
Statistical Analysis 1: Comparison: PK-Driven Prophylaxis vs Standard Prophylaxis; Test type: Superiority or Other; p = 0.1467, Wilcoxon-Rank Sum (Mann-Whitney)

27. Secondary Outcome: Bodily Pain HRQoL Scores Change From On-Demand Period Through Prophylaxis Period
Description: Change = (End of on-demand treatment) - (End of prophylaxis regimen). A negative value for the median difference equates to a larger domain score for the prophylaxis regimen. Scores range 0-100, higher scores represent better health. There is no total overall score; scoring is done for subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores.
Time Frame: End of on-demand treatment period (6 months) and at study termination (approximately 18 months)
Population: Pharmacoeconomic analysis set for participants ≥14 years of age
Measure: Median (Full Range); unit: Scores on a scale
Groups:
- ≥14 Years of Age: After an on-demand treatment period, participants were randomized to 1 of 2 prophylactic regimens for 12 months. The standard prophylactic regimen was dosed at 20 to 40 IU/kg every 48 ±6 hours, and the PK-driven prophylaxis regimen was dosed at 20 to 80 IU/kg every 72 ±6 hours.
Arm/Group | ≥14 Years of Age
Number analyzed (Participants) | 57
Scores on a scale | 0.00 [-29.55 to 17.55]
Statistical Analysis 1: Comparison: ≥14 Years of Age; Test type: Superiority or Other; p = 0.0007, Wilcoxon signed-rank test — Due to multiple hypotheses testing results, adjusted alpha values are set to α*=0.005 (0.05/10). Adjustments take into account 10 hypotheses tests between On-Demand and any Prophylaxis. Statistically significant results are considered p-values < α*

28. Secondary Outcome: Physical Component Scores (PCS) HRQoL Scores Change From On-Demand Period Through Prophylaxis Period
Description: Change = (End of on-demand treatment) - (End of prophylaxis regimen) A negative value for the median difference equates to a larger domain score for the prophylaxis regimen. Scores range 0-100, higher scores represent better health. There is no total overall score; scoring is done for subscores and summary scores. The raw data from the SF-36 items were transformed to norm based scores.
Time Frame: End of on-demand treatment period (6 months) and at study termination (approximately 18 months)
Population: Pharmacoeconomic analysis set for participants ≥14 years of age
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | ≥14 Years of Age
Number analyzed (Participants) | 57
Scores on a scale | -2.76 [-20.22 to 19.70]
Statistical Analysis 1: Comparison: ≥14 Years of Age; Test type: Superiority or Other; p = 0.0002, Wilcoxon signed-rank test — [p-value comment as in outcome 27, analysis 1]

29. Post Hoc Outcome: Median (IQR) Annualized Bleed Rates
Description: Bleed rates (number of bleeding episodes per subject) were annualized to account for the varying number of days a subject may have actually been on each regimen.
Time Frame: On-demand 6 months (± 2 weeks); Prophylaxis 12 months (± 2 weeks)
Population: Per-Protocol Efficacy Analysis Set
Measure: Median (Inter-Quartile Range); unit: Bleeding episodes
Groups:
- On-Demand Regimen: After the initial PK study, a 6 month period of on-demand treatment was conducted (Part 1)
- Standard Prophylaxis: Dosed at 20 to 40 IU/kg every 48 ±6 hours for 12 months (Part 2)
- PK-driven Prophylaxis: Dosed at 20 to 80 IU/kg every 72 ±6 hours for 12 months (Part 2)
- Any Prophylaxis: Either Standard or PK-driven Prophylaxis
Arm/Group | On-Demand Regimen | Standard Prophylaxis | PK-driven Prophylaxis | Any Prophylaxis
Number analyzed (Participants) | 53 | 30 | 23 | 53
Bleeding episodes | 43.98 [35.73 to 56.53] | 0.99 [0.00 to 2.14] | 1.00 [0.00 to 4.08] | 1.00 [0.00 to 4.07]
Statistical Analysis 1: Comparison: On-Demand Regimen vs Any Prophylaxis; Test type: Superiority or Other; p < 0.0001, Wilcoxon Signed-Rank Test

ADVERSE EVENTS:
Time Frame: Throughout the study period (4 years and 5 months)
Groups:
- On-Demand: On-demand: rAHF-PFM was to be used for the treatment of bleeding episodes according to the severity and type of episode by the protocol-recommended dosing until the episode resolved: superficial (10-20 IU/kg every 12-14 hours), minor joint (20-40 IU/kg every 12-14 hours), deep muscle (30-60 IU/kg every 12-14 hours), major joint or life-threatening (60-100 IU/kg every 8-12 hours), genitourinary, GI, and intracranial (60-100 IU/kg every 8-12 hours)
- Standard Prophylaxis: Standard prophylaxis regimen dosed at 20 to 40 IU/kg (every 48 ±6 hours), exact regimen to be determined by the investigator
- PK-Driven Prophylaxis: PK-driven prophylaxis regimen dosed at 20 to 80 IU/kg (every 72 ±6 hours) exact regimen to be determined by the sponsor
Arm/Group | On-Demand | Standard Prophylaxis | PK-Driven Prophylaxis | SAEs Outside of the 3 Treatment Arms
Serious Adverse Events (participants affected / at risk) | 7/73 | 2/32 | 3/34 | 1/1
Other Adverse Events (participants affected / at risk) | 18/73 | 4/32 | 7/34 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-Demand (N=73) | Standard Prophylaxis (N=32) | PK-Driven Prophylaxis (N=34) | SAEs Outside of the 3 Treatment Arms (N=1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMOPHILIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOSPITALIZATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULPITIS DENTAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SOMNAMBULISM (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACTOR VIII INHIBITION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — This event was unconfirmed and therefore did not meet protocol definition for a Factor VIII inhibitor.
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-Demand (N=73) | Standard Prophylaxis (N=32) | PK-Driven Prophylaxis (N=34) | SAEs Outside of the 3 Treatment Arms (N=1)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (6) | 0 (0) | 3 (5) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or ≤2 years after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥60 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., intellectual property protection)